CLINICAL TRIAL: NCT02434887
Title: Clinical Study for Perceived Effectiveness Evaluation of Moisturizing Action of Intimate Use Product in Postmenopausal Women
Acronym: CLIN ST EF EV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kley Hertz S/A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: KLEY HERTZ-004
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Female Dry Genital Mucosa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: KL029 Intimate Lubricant Gel

INTERVENTIONS:
Device: KL029 Intimate Lubricant Gel

SUMMARY:
The purpose of this study is to verify the effectiveness of the investigational product through Subjective Assessment and answered by volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Female aged between 45 to 65 years old
* Sexually active volunteers, with a minimum of 1 intercourse per week
* In menopause for at least 6 months;
* Intact skin in the product analysis region;
* No prior reactions to topical products
* Reading, understanding, agreement and signature of the informed consent form

Exclusion Criteria:

* Use of anti-inflammatory and immunosuppressive ( in the last 30 days and during the study)
* Active skin diseases (local or disseminated) in the evaluation área;
* Diseases that cause imune suppression;
* Endocrine disorders such as thyroid, ovarian or adrenal gland disorders;
* Any infection in the region where the product will be analyzed diagnosed at enrollment;
* Other conditions considered by the investigator physician as reasonable for the disqualification of the individual's participation in the study.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of the product's efficiency as a moisturizer through subjective evaluation | 40 days